CLINICAL TRIAL: NCT05578521
Title: CerebrAlcare Pills on CereBral Small VesseL DiseasE（CABLE）：A Randomized, Double-blinded, Placebo-controlled, Multi-center Trial
Brief Title: CerebrAlcare Pills on CereBral Small VesseL DiseasE（CABLE）
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY-2021-176-04
Record Dates: First submitted 2022-07-24; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: cerebral small vessel diseases; Cerebralcare Pills; cognitive function; randomized controlled trial; multicenter study; double blind study; placebo-controlled
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebralcare pills placebo group (Placebo Comparator): This group will receive Cerebralcare pills placebo, 2 packages, twice a day, from the day of randomization to 6 months.
  Interventions: Drug: Cerebralcare pills placebo
- Cerebralcare pills group (Experimental): This group will receive Cerebralcare pills, 2 packages, twice a day, from the day of randomization to 6 months.
  Interventions: Drug: Cerebralcare pills

INTERVENTIONS:
Drug: Cerebralcare pills — a dose of 2 packages, twice a day of Cerebralcare pills
  Arms: Cerebralcare pills group
Drug: Cerebralcare pills placebo — Cerebralcare pills placebo will be administrated at the same rate with experimental group
  Arms: Cerebralcare pills placebo group

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multicenter trial. Cerebral small vessel disease (CSVD) patients will be diagnosed by Magnetic Resonance Imaging (MRI) and randomized into treatment or control groups. The purpose of this trial is to assess the efficacy of cerebralcare pills on cerebral small vessel disease.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) is prevalent in the aging population with insidious onset, almost affecting all levels of the brain vasculature, and challenges the social and healthcare system worldwide. CSVD is the major cause of 25% of strokes and more than doubles the odds of recurrent stroke; furthermore, it contributes to 45% of dementia cases and to global functional decline. However, an incomplete understanding of the pathogenesis of CSVD limits prevention and treatment efforts.

Cerebralcare Granule (CG) or Yangxue Qingnao granule, is a polyherbal medicine that was approved in 1997 by the China State Food and Drug Administration for the treatment of headaches and dizziness associated with cerebrovascular diseases. Cerebralcare pill is composed of 11 herbs. These herbs contain small molecules with various pharmacological actions. Cerebralcare pills have the same component as CG. Previous studies have demonstrated that CG significantly attenuated ischemia-reperfusion induced dysfunction, structural abnormalities in the microcirculation, and inflammatory injury. There are also studies confirming that CG also improved cognition function, improved cerebral microcirculation disorders, and hemodynamics.

Patients enrolled will be randomly assigned to either the treatment or control group to receive Brain Pill/Brain Pill placebo (from randomization to 6 months at a dose of 2 packs per day). Face-to-face interviews will be conducted at baseline, day 90, day 180, and 1 year after randomization.

The primary endpoint is the progression in cognition function which is assessed by Montreal Cognitive Assessment (MoCA) score. The secondary endpoints include changes in clinical characters, imaging markers (number and volume of white matter, number of lacunes, microbleeds, enlarged perivascular space ), hemodynamic parameters, Chinese medical symptoms, blood-brain barrier (BBB) permeability, proteomics, and inflammatory markers. The safety endpoints include severe hemorrhage events, symptomatic and asymptomatic intracranial hemorrhage, moderate hemorrhage, overall mortality, and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. 45-75 years old;
2. No gender limitation;
3. Cerebral small vessel disease is observed on brain MRI. White matter hyperintensity, Fazekas score ≥ 1 and combined more than 2 vascular risk factors (hypertension, hyperlipidemia, diabetes, obesity, smoking, and other vascular events except stroke) or combined with lacunar focus or Imaging findings suggest new subcortical lacunar infarction (within 7 days).
4. Mild or moderate vascular cognitive impairment(16 ≤ MoCA ≤ 24 score, for patients with primary school degree or below,15 ≤ MoCA ≤ 23 score).
5. Daily life independence (mRS ≤ 2).
6. Sign informed consent.

Note:

1. The imaging definition of small vessel disease refers to the strong guideline The total score of Fazekas was 6, which was the sum of Fazekas scores of subcortical and periventricular white matter lesions.
2. New subcortical lacunar infarction: head MRI examination, subcortical, basal ganglia or brain stem DWI showed high signal (ADC diffusion limited) lesions with diameter < 20 mm, with or without corresponding clinical symptoms; There were new clinical symptoms. FLAIR sequence of head MRI showed flair hyperintense lesions (diameter < 20 mm) in subcortical, basal ganglia or pons.

Exclusion Criteria:

1. Cerebral hemorrhage and subarachnoid hemorrhage occurred within 30 days.
2. Symptomatic middle cerebral artery and/or internal carotid artery stenosis, stenosis rate ≥ 50%; asymptomatic middle cerebral artery and/or internal carotid artery stenosis, stenosis rate ≥ 70%.
3. Coronary CTA or coronary angiography showed severe three vessel lesions or frequent angina pectoris within 30 days.
4. Chronic kidney disease stage 4 or 5.
5. Resistant hypertension which could not be controlled by medicine (SBP > 180mmHg or DBP > 110mmHg).
6. Resistant hyperglycemia which could not be controlled by medicine（fasting blood glucose > 10mmol/L or HB1AC > 7%).
7. In acute cerebral infarction, the lesions showed high signal intensity on DWI, and the diameter was more than 20 mm or history of assive cerebral infarction within 30 days.
8. Neurodegenerative diseases, such as AD and PD, have been diagnosed.
9. There are clear non angiogenic white matter lesions, such as multiple sclerosis, adult white matter dysplasia, metabolic encephalopathy diseases, etc.
10. Untreated cerebrovascular malformations or intracranial aneurysms (d > 3mm).
11. Active gastrointestinal bleeding.
12. Coagulation dysfunction or history of systemic bleeding.
13. Hemorrhagic tendency (including but not limited to)：PLT<100×109/L; heparin treatment within 48h; APTT ≥ 35s; current use of warfarin, INR > 1.7; current use of novel oral anticoagulants; current use of direct thrombin or factor Xa inhibitor.
14. Severe hepatic or renal or heat insufficiency before randomization (severe hepatic insufficiency refers to ALT or AST > 2 times the upper limit of normal; severe renal insufficiency refers to serum creatinine> 1.5 times the upper limit of normal or eGFR<40 ml/min/1.73m2; severe heat insufficiency refers to NYHA stage 3 and 4).
15. History of intracranial or intramedullary surgery within three months of randomization.
16. The patient has used or is using chinese medicine with similar components to CerebrAlcare pill/granule (including Tianshu capsule, Toutongning capsule, Naoxintong capsule, Danzhen Toutou capsule, Yindanxinnaotong soft capsule, Naoxinqing Tablet, Bazhen pill and Shiquandabu pill) within 14 days.
17. Definite indications for anticoagulation (suspicion of cardioembolism, e.g. atrial fibrillation, known heart valve prosthesis, atrial myxoma, endocarditis, etc.) or definite indications for dual antiplatelet therapy (e.g. recent coronary or cerebral artery stent implantation).
18. Other surgical or interventional therapy planned within 1 year requiring experimental drugs discontinuation.
19. Childbearing-age women who do not take effective methods of contraception without negative records of pregnancy tests.
20. Known to be allergic to CerebrAlcare pill/granule.
21. Contraindications of MRI examination (such as claustrophobia).
22. With severe organic diseases, such as malignant tumor, the expected survival time is less than 1 years.
23. Due to geographical or other reasons can not cooperate to complete the follow-up.
24. Patients also participated in other clinical trials.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression in cognition function | 6 months after randomization
  Cognition function assessed by Montreal Cognitive Assessment (MoCA) score. Score range 0-30. Higher scores mean a better outcome..

SECONDARY OUTCOMES:
Changes in both systolic and diastolic blood pressure | 3 months, 6 months and 1 year after randomization
  Including systolic and diastolic blood pressure (mmHg).
Rey auditory verbal learning test（RAVLT） | 3 months, 6 months and 1 year after randomization
  The Rey Auditory Verbal Learning Test (RAVLT) provides a standardized procedure to evaluate a range of aspects of verbal learning and memory of supra-span lists of words. The test requires recalling as many words as possible in any order from a standard list of 15 unrelated words read out by the examiner. The total score ranges from 0-120, with a lower score indicating a worse outcome.
Generalized Anxiety Disorder 7（GAD-7) | 3 months, 6 months and 1 year after randomization
  Generalized Anxiety disorder (GAD) is a widespread psychiatric syndrome involving significant consequences on people's health, with a total score of 21, where a higher score means a worse outcome. However, recent data show that this disorder has received little attention when compared to other anxiety disorders.
Self-rating depression scale | 3 months, 6 months and 1 year after randomization
  The Zung Self-Rating Depression Scale (SDS) consists of 20 items with a Likert type scale after each item. Each item is rated from 1 to 4, with scores ranging from 20 to 80, where higher scores mean worse results
Dizziness handicap inventory（DHI） | 3 months, 6 months and 1 year after randomization
  The DHI has 25 items with 3 response levels, sub-grouped into three domains: functional, emotional, and physical. A shortened version, the Dizziness Handicap Inventory short form (DHIsf), reduced to 13 items with 2 response levels, has been shown to compare favourably to the original version. Scores range from 0-100, with higher scores indicating worse outcomes.
Headache impact test 6(HIT-6） | 3 months, 6 months and 1 year after randomization
  The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress.Total HIT-6 score that ranges from 36 to 78, where a lower score indicates a greater impact of headache on the daily life of the respondent.
EuroQol five dimensions questionnaire (EQ-5D) | 3 months, 6 months and 1 year after randomization
  It includes a descriptive system(DS) and a visual analogue scale(VAS). Two indicators are index value(ranged 0-1) and visual score(ranged 0-100) with higher scores corresponding to better health status.
Stroop Color Word Test | 3 months, 6 months and 1 year after randomization
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. Shorter the test time, the better the outcome.
Severity of white matter hyperintensities(WMHs) | 6 months and 1 year after randomization
  Fazekas score is used to describe the different types of hyperintense signal abnormalities surrounding the ventricles and in the deep white matter. Periventricular hyperintensity (PVH) is graded as 0 = absence, 1 = "caps" or pencil-thin lining, 2 = smooth "halo", 3 = irregular PVH extending into the deep white matter. Separate deep white matter hyperintensity (DWMH) is rated as 0 = absence, 1 = punctate foci, 2 = beginning confluence of foci, 3 = large confluent areas. Higher scores indicats a worse outcome.
Changes of white matter hyperintensities(WMHs) volume | 6 months and 1 year after randomization
  WMH volume is assessed on 3D fluid attenuated inversion recovery (FLAIR) sequence in mm3 or cm3. Larger volume indicates a worse outcome.
Number of lacunes | 6 months and 1 year after randomization
  Lacunes were defined as rounded or ovoid lesions in the subcortical, basal ganglia, or brainstem, ranging from 3mm to 20mm in diameter, presenting with cerebral spinal fluid signal intensity on T2 and FLAIR, generally featuring a hyperintense rim on FLAIR and no increased signal on diffusion weighted imaging (DWI). Higher number of lacunae means a worse outcome.
Number of cerebral microbleeds | 6 months and 1 year after randomization
  Cerebral microbleeds are defined as rounded, hypodense foci within brain parenchyma on susceptibi lity weighted imaging (SWI) sequence, up to 10 mm in diameter, and were differentiated from microbleed mimics based on current guidelines. Higher number of cerebral microbleeds means a worse outcome.
Number of enlarged perivascular space | 6 months and 1 year after randomization
  Enlarged perivascular space was defined as small punctate or linear hyperintensities on T2 images in the basal ganglia or centrum semiovale. Higher number of enlarged perivascular spaces means a worse outcome.
Changes in hemodynamic parameters | 6 months and 1 year after randomization
  Lower cerebrovascular reactivity (CVR), cerebral blood flow (CBF), and reduced radial peripapillary capillary network density, and parafoveal vessel densities of the superficial retinal capillary plexuses mean worse outcomes.
changes in Chinese medical symptoms | 6 months and 1 year after randomization
  Chinese medical symptoms assessed by Blood Deficiency and Liver Hyperactivity Syndrome score. Scores range 0-21 and higher scores mean a worse outcome.
Difference of recurrent stroke between groups | 3 months, 6 months and 1 year after randomization
  stroke included ischemic stroke, hemorrhagic stroke, TIA, et al.
changes in Blood-Brain Barrier (BBB) Permeability between groups | 6 months and 1 year after randomization
  BBB permeability is assessed by MRI and biomarker (including NSE, GFAP, S100β).
Compare protein profiles observed among different groups. | 6 months and 1 year after randomization
  Blood was collected from the healthy (n=6), experimental (n=6) and placebo (n=6) groups at baseline, 3 months, and 12 months post-dosing. Alterations in protein profiles were detected by high performance liquid chromatography-mass spectrometry (HPLC-MS). GO classification and pathway enrichment were performed to analyse relevant protein changes. Serum metabolomics was determined using untargeted assays, and metabolite patterns in different groups were distinguished using orthogonal partial least squares analysis (OPLS-DA), compared with databases, and validated with the help of standards to finalise qualitative and quantitative analysis of metabolites and to identify differential metabolites. The Cell Counting Bead Analysis (CBA) Flex Set Flow Multifactor Assay Kit is used to detect serum levels of the inflammatory factors IL-1β, IL-6, IL-10, IL-12 and TNF-α. Western blot analysis is used to validate changes in the expression of 20 key proteins obtained from proteomic analysis.
Composite vascular events | 3 months, 6 months and 1 year after randomization
  Incidence of symptomatic stroke, myocardial infarction and vascular death.
All-cause death | 3 months, 6 months and 1 year after randomization
  Deaths from all causes to the research subjects
Moderate and/or severe hemorrhage events | 3 months, 6 months and 1 year after randomization
  According to Global Utilization of Streptokinase and t-PA for Occluded Coronary Arteries (GUSTO) criteria which classifies the severity of bleeding complications as follows: 1) severe or life-threatening bleeding-intracranial bleeding or bleeding that causes substantial hemodynamic compromise requiring treatment; 2) moderate bleeding-bleeding which needs blood transfusion; 3) minor bleeding-other bleeding, neither requiring transfusion nor causing hemodynamic compromise.
Symptomatic and/or asymptomatic intracranial hemorrhage | 3 months, 6 months and 1 year after randomization
Adverse events and severe adverse events | 3 months, 6 months and 1 year after randomization
  renal failure, hepatic failure, death.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD，MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou M, Gong Y, Han S, Wang M, Gu W, Chen HS, Zheng W, Feng K, Wang D, Li H, Zheng Z, Pan Y, Chen W, Wang Y. CerebrAlcare Pills on CereBral Small VesseL DiseasE (CABLE) trial: rationale and design. Stroke Vasc Neurol. 2025 Sep 2:svn-2024-003756. doi: 10.1136/svn-2024-003756. Online ahead of print. PMID 40897453